CLINICAL TRIAL: NCT07194902
Title: HIV Self-testing for Partners of HIV-uninfected Postpartum Women to Facilitate PrEP and Antiretroviral Therapy Uptake to Promote HIV Treatment and Prevention
Brief Title: HIV Self-testing for Partners of HIV-uninfected Postpartum Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christina Psaros, Associate Director, Behavioral Medicine, Department of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025P002271; R34MH132446 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HIV Self-testing; Male Partners of HIV-negative Postpartum Women; PrEP Uptake; Feasibility; Acceptability; HIV Prevention
Keywords: HIV Prevention; PrEP; HIV Self-Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- H4P Intervention Arm (Active Comparator): At one of their last scheduled antenatal care visits (i.e., between 30- 40 weeks' gestation), all female participants will be provided with up to three HIVST kits for male partner distribution, and will be provided with information and a demonstration per the standard of care (SOC) for HIVST kit distribution. In addition to what female participants in the control arm engage in, they will engage in 30-45 minutes HIVST and PrEP uptake counseling intervention at the baseline visit. Male partners, in addition to the SOC written information provided to the control arm, will also receive a QR code linked to a brief video created by the study team. The video will communicate, among other things, information on geographically diverse HIV treatment resources, and why linkage to HIV care is needed in the context of the relationship (e.g., increased risk for HIV during the postpartum period, risk of transmission to infant during breastfeeding, his role in protecting the family's health).
  Interventions: Behavioral: HIVST for Partners and PrEP uptake for HIV-uninfected Postpartum Women ("H4P").
- Control Arm (Placebo Comparator): At one of their last scheduled antenatal care visits (i.e., between 30- 40 weeks' gestation), all female participants will be provided with up to three HIVST kits for male partner distribution, and will receive 15-20 minutes of counseling. Female participants will receive OraQuick Rapid HIV-1/2 Antibody Tests. OraQuick kits will include step-by-step instructions on use and interpretation of results. All female participants will be provided with information and a demonstration per the standard of care (SOC) for HIVST kit distribution and will engage in a brief exercise that involves evaluating the pros and cons of offering HIVST kits to their partners. All men will be provided with the HIVST kit by their female partners (including directions for use, consistent with SOC), along with a letter describing how to contact the study team.
  Interventions: Behavioral: HIVST for Partners and PrEP uptake for HIV-uninfected Postpartum Women ("H4P").

INTERVENTIONS:
Behavioral: HIVST for Partners and PrEP uptake for HIV-uninfected Postpartum Women ("H4P"). — For female participants, the intervention includes a 30-45 minute counseling session that will cover (1) SOC PrEP information, (2) communications skills training for HIVST kit distribution, (3) Motivational interviewing strategies (e.g., PrEP/HIVST pros/cons), (4) problem-solving barriers to PrEP uptake or HIVST distribution, (5) linkage enablers (e.g., care sites, transportation, asking questions of providers). For their male partners, an informative video will cover geographically diverse HIV treatment resources, as well as on why linkage to HIV care is needed in the context of the relationship with his female partner and gender norms. The video will also demonstrate a brief motivational exercise whereby men are asked to consider the pros and cons of linking to HIV care versus not (with examples), as well as a step-by-step guide to generate a concrete plan for linkage to care based on "linkage enablers".

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of a combination intervention to promote HIV self-testing (HIVST) for Partners and PrEP uptake for HIV-uninfected Postpartum Women ("H4P"). H4P includes evidence-based cognitive behavioral therapy (CBT) strategies, such as communication skills training, motivational interviewing, and problem-solving. The investigators will conduct a randomized pilot trial of the H4P intervention to evaluate the feasibility, acceptability, and preliminary effectiveness of a multi-step PrEP uptake and HIV self-test kit intervention for postpartum HIV-uninfected women (N = 60 and their male partners) who report a partner of unknown serostatus, and their partners, in the province of KwaZulu-Natal, South Africa.

ELIGIBILITY:
Female Inclusion Criteria:

* woman
* Age ≥18
* ≥30 weeks pregnant per medical record due date
* non-reactive third trimester HIV test (verified from their antenatal care chart)
* reporting at least one unknown-serostatus partner
* fluent in English or isiZulu
* willing to give researchers permission to contact them for repeated assessments
* able to provide informed consent

Male Inclusion Criteria: partners meeting the inclusion criteria as described above, and who complete verification questions to confirm their identity and status as the partners of the enrolled female participants. Additional inclusion criteria for men include:

* man
* Age ≥18
* partner of enrolled women, confirmed via couples verification tool
* fluent in English or isiZulu
* willing to give researchers permission to contact them
* able to provide informed consent.

Exclusion Criteria: Individuals with significant psychiatric illness that could interfere with participation or the ability to provide informed consent will be excluded at the discretion of the study team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention | Baseline and 3-month follow-up
  To evaluate feasibility, the investigators will examine and report on (1) the number of participants (female and male) screened, eligible, and enrolled (whether > 70% of those screened enroll/agree to participate); (2) the number of female participants who distribute a kit to their male partner; the number of female participants who learn their male partner's status; and the number of male partners who use the kit, complete HIVST verification, use the QR code, and complete confirmatory testing.
Acceptability | Post-Intervention
  Acceptability will be evaluated using the Client Satisfaction Questionnaire (CSQ8). The investigators will also record data on reasons for declining enrollment, and will document failure to distribute or use the kit, complete verification, and complete confirmatory testing. All qualitative exit interview data will be explored for categories and themes around intervention acceptability. Qualitative data will be analyzed using content analysis, an iterative, multi-step process as described by Miles and Huberman and Strauss and Corbin.
Safety concerns as a result of HIVST distribution | Baseline and 3-month follow-up
  Safety will be evaluated via self-report of any safety concerns anticipated or experienced as a result of HIVST distribution including social, emotional, or physical harms. Female participants will be screened for partner violence (Abuse Assessment Screen) at baseline. If female participants report being a victim of violence, study staff will contact the local site PI/Co-PI (Smit/Mosery) and an appropriate clinical intervention will be delivered. Participants with elevated scores will be provided with a referral for mental health services, using referral systems that are already in place in Dr. Psaros' R01 (R01MH112385) and will be asked to not distribute the kits but stay in the study, as they might benefit from the intervention session. This will also be explored in qualitative interviews (as described above).
Preliminary effectiveness of H4P intervention. | 3-month follow-up
  Women: Preliminary effectiveness: Proportion of women whose male partners test positive or do not test/share result who initiate and use PrEP at 3 months postpartum, via self-report, and point of care test for tenofovir, via urine dipstick test which reflects use in the past few days.
  Men: Preliminary effectiveness: Proportion of men with a positive test who link to care, via self-report and paper test result or CD4/viral load result from confirmatory testing, and copy of treatment regimen (or photographs of these documents).
Challenges, successes, barriers, facilitators, and preferences for optimizing H4P intervention. | 3-month follow-up
  Qualitative exit interviews: Conducted with subsets of women and men assigned to the H4P intervention arm (based on HIV self-test kit distribution, kit use, and linkage) to explore challenges (including gender-based violence), successes, barriers (e.g., motivation to test for HIV during the postpartum period for men), facilitators, preferences around HIV self-test kit distribution (including use of Quick Response codes), HIV self-testing verification, confirmatory testing and verification, and linkage to care (e.g., PrEP or Antiretroviral Therapy, including how women decided to initiate PrEP, and experiences with PrEP linkage and clinic support around PrEP use), and opportunities to optimize the H4P intervention.

SECONDARY OUTCOMES:
Estimate PrEP uptake among female participants | 3-month follow-up
  The investigators will estimate PrEP uptake among female participants in a separate logistic regression model, adjusting for covariates carefully given the feasibility/acceptability design and small N.
HIV and Pregnancy characteristics | Baseline and 3-month follow-up
  Women: Results of HIV tests (3-month follow-up only); gravity, parity, number of weeks gestation when enrolled in Antenatal Care, ever offered PrEP, ever used PrEP, ever completed couples based counseling and testing. Pregnancy intention: Pregnancy Risk Assessment Monitoring System survey: Up to 4 items assessing attitudes and feelings about the most recent pregnancy.
  Men: Date of last HIV test, ever completed couples-based counseling and testing, history of prior positive test (and date), whether currently taking Antiretroviral Therapy, and number of children. Referent pregnancy intention: Pregnancy Risk Assessment Monitoring System survey.
Physical health | Baseline and 3-month follow-up
  Multi-Country Study on Women's Health and Violence Core Questionnaire Version 9: 43-item General Health section to measure overall health status and physical symptoms.
Depression | Baseline and 3-month follow-up
  Women: Edinburgh Postnatal Depression Scale: 10-item scale widely used and validated in South Africa among both pregnant and postpartum women.
  Men: Center for Epidemiologic Studies Depression scale: 20-item measure of depressive symptoms. High internal consistency; widely used in South Africa.
Substance Use | Baseline and 3-month follow-up
  Addiction Severity Index-Lite: Assesses lifetime and recent substance use, including severity. Up to 111 items; previously used in South Africa.
Health beliefs | Baseline
  Women: Perceived Risk of HIV Infection Scale: 8-item measure of how people perceive their personal risk of HIV. Validated with women in Sub-Saharan Africa. PrEP Optimism: 3 items to assess beliefs about PrEP efficacy in preventing HIV. Items used among HIV-uninfected pregnant women and heterosexual couples in South Africa. Men: Antiretroviral Therapy treatment beliefs: Beliefs about Medicines Questionnaire: Two five-item scales assessing beliefs about the necessity of and concerns about taking prescribed medication. Used in Sub-Saharan Africa.
Relationship characteristics and communication | Baseline and 3-month follow-up
  Partner Communication Scale: 5-item measure of sexual communication between partners around condom use, HIV/STI prevention, pregnancy, and sexual history. Internal consistency has been established. Dyadic Trust Scale: 8- item measures of trust in close relationships. Used and validated in South Africa and other resource-limited settings. Gender-Equitable Men Scale: 24-item measure of attitudes towards gender relations. Used and validated among women in South Africa and other resource-limited settings. Sexual Relationship Power Scale: 23-item measure of decision-making dominance and relationship control. Validated among women in South Africa. Duration of relationship will be assessed.
Partner Violence | Baseline and 3-month follow-up
  Women: Abuse Assessment Screen: 5-item measure of presence of violence in the last year. Clinical assessment conducted if answer is "yes" to ≥1 questions. Widely used among those who are pregnant and validated among pregnant women in resource-limited settings
HIV-related stigma | Baseline and 3-month follow-up
  Personal Stigma and Attributed Stigma Scales: parallel 17-item scales to measure personal stigmatizing views about HIV and stigma attributed to others. Both scales validated among HIV-uninfected women in South Africa.
  PrEP Use Stigma Scale: 6-item scale measuring internalized stigma related to HIV and PrEP use, adapted for use among young women in Zimbabwe and South Africa (Cronbach's alpha: 0.89).
Structural barriers | Baseline and 3-month follow-up
  Modes and costs of transportation to travel to clinic, travel time to clinic visits, and the average amount of time spent at the clinic.
Demographics | Baseline
  Age; ethnicity; country of origin; educational level; employment status; occupation; income; religion; housing stability; with whom participant lives.

CONTACTS AND LOCATIONS:
Locations (1):
- Wits MatCH Research Unit, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Undecided